CLINICAL TRIAL: NCT02508675
Title: Prevalence, Recovery Patterns and Risk Factors of Non-fatal Outcome and Costs After Trauma; a Prospective Follow up Study
Brief Title: Non-fatal Outcome After Trauma
Acronym: βioς
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Network Emergency Care Brabant (Other)
Collaborators: Elisabeth-TweeSteden Ziekenhuis (Other); Erasmus Medical Center (Other); Tilburg University (Other); Amphia Hospital (Other); Catharina Ziekenhuis Eindhoven (Other); Bravis Hospital (Other); Elkerliek Hospital (Other); Maas Hospital Pantein (Other); St. Anna Ziekenhuis, Geldrop, Netherlands (Other); Jeroen Bosch Ziekenhuis (Other); Maxima Medical Center (Other); Twee Steden Hospital (Unknown); Bernhoven Hospital (Other); Maasstad Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NL50258.028.14
Record Dates: First submitted 2015-07-23; First posted 2015-07-27 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Trauma
Keywords: injury; risk factors; outcome; costs
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The major aim of this project is to investigate the prevalence, recovery patterns and risk factors for health related quality of life functional, psychological, societal and economic outcome after trauma. Another aim is to validate the WHO Quality Of Life-bref (WHOQOL-Bref) questionnaire for the trauma population.

DETAILED DESCRIPTION:
Patients aged 18 years and older admitted in a hospital in Brabant after a trauma, independent of severity or type of injury are included in the study. Patients who decease during hospital stay or transferred to another hospital outside the borders of trauma region Brabant will be excluded. Socio-demographic characteristics, functional and psychological outcome and Health Related Quality of Life (HRQoL) shortly after trauma will be measured. Subsequently the same items will be measured after 1, 3, 6, 12 and 24 months. Outcomes will be assessed using questionnaires. The primary outcome parameters are: short and long term HRQoL, functional and psychological outcome, and Healthcare and societal costs in injured patients. Secondary outcome measures are Return to Work and health care consumption.

ELIGIBILITY:
Inclusion Criteria:

* patients seen at the ED which are admitted to the ICU or ward after getting injured
* all types and severities of injury (Injury Severity Score (ISS) 1-75)
* a minimal age of 18 years old
* sufficient knowledge of the Dutch language

Exclusion Criteria:

* patients who are dead on arrival or decease in the ED
* pathological fracture (i.e., the bones are weakened by disease, for example by a tumor)
* patients who die in the hospital will drop out the study and will not be included in the analyses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients seen at the Emergency Department (ED) which are admitted to the Intensive Care Unit (ICU) or ward after getting injured, with a minimal age of 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 6500 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Short and longterm HRQoL | 2 years
  self-reported questionnaire
Functional outcome | 2 years
  self-reported questionnaire
Healthcare and societal costs | 2 years
  self-reported questionnaire and information from registries
Psychological outcome | 2 years
  self-reported questionnaire
Social outcome | 2 years
  self-reported questionnaire

SECONDARY OUTCOMES:
Return to work (RtW) | 2 years
  self-reported questionnaire
Health care consumption | 2 years
  self-reported questionnaire and information from registries

CONTACTS AND LOCATIONS:
Overall Officials: Koen W Lansink, MD, Principal Investigator — St. Elisabeth Hospital, Tilburg, The Netherlands; Mariska A de Jongh, PhD, Principal Investigator — Network Emergency Care Brabant

REFERENCES:
- [Derived] de Munter L, van de Ree CLP, van der Jagt OP, Gosens T, Maas HAAM, de Jongh MAC. Trajectories and prognostic factors for recovery after hip fracture: a longitudinal cohort study. Int Orthop. 2022 Dec;46(12):2913-2926. doi: 10.1007/s00264-022-05561-4. Epub 2022 Sep 6. PMID 36066616
- [Derived] de Munter L, Polinder S, Havermans RJM, Steyerberg EW, de Jongh MAC. Prognostic factors for recovery of health status after injury: a prospective multicentre cohort study. BMJ Open. 2021 Jan 6;11(1):e038707. doi: 10.1136/bmjopen-2020-038707. PMID 33408198
- [Derived] Brouwers L, de Jongh MAC, de Munter L, Edwards M, Lansink KWW. Prognostic factors and quality of life after pelvic fractures. The Brabant Injury Outcome Surveillance (BIOS) study. PLoS One. 2020 Jun 11;15(6):e0233690. doi: 10.1371/journal.pone.0233690. eCollection 2020. PMID 32525901
- [Derived] Kruithof N, Polinder S, de Munter L, van de Ree CLP, Lansink KWW, de Jongh MAC; BIOS-group. Health status and psychological outcomes after trauma: A prospective multicenter cohort study. PLoS One. 2020 Apr 21;15(4):e0231649. doi: 10.1371/journal.pone.0231649. eCollection 2020. PMID 32315373
- [Derived] de Munter L, Polinder S, Haagsma JA, Kruithof N, van de Ree CLP, Steyerberg EW, de Jongh M. Prevalence and Prognostic Factors for Psychological Distress After Trauma. Arch Phys Med Rehabil. 2020 May;101(5):877-884. doi: 10.1016/j.apmr.2019.10.196. Epub 2019 Dec 23. PMID 31874154
- [Derived] van de Ree CLP, Landers MJF, Kruithof N, de Munter L, Slaets JPJ, Gosens T, de Jongh MAC. Effect of frailty on quality of life in elderly patients after hip fracture: a longitudinal study. BMJ Open. 2019 Jul 18;9(7):e025941. doi: 10.1136/bmjopen-2018-025941. PMID 31324679
- [Derived] Kruithof N, Haagsma JA, Karabatzakis M, Cnossen MC, de Munter L, van de Ree CLP, de Jongh MAC, Polinder S. Validation and reliability of the Abbreviated World Health Organization Quality of Life Instrument (WHOQOL-BREF) in the hospitalized trauma population. Injury. 2018 Oct;49(10):1796-1804. doi: 10.1016/j.injury.2018.08.016. Epub 2018 Aug 23. PMID 30154022
- [Derived] de Jongh MA, Kruithof N, Gosens T, van de Ree CL, de Munter L, Brouwers L, Polinder S, Lansink KW; BIOS-group. Prevalence, recovery patterns and predictors of quality of life and costs after non-fatal injury: the Brabant Injury Outcome Surveillance (BIOS) study. Inj Prev. 2017 Feb;23(1):59. doi: 10.1136/injuryprev-2016-042032. Epub 2016 May 6. PMID 27154507